CLINICAL TRIAL: NCT06024187
Title: Necrosis After Cold Dissection Versus Electrocautery Dissection in Endoscopic Nipple-Sparing Mastectomy and Immediate Implant-Based Reconstruction: A Prospective Randomized Controlled Trial
Brief Title: Cold Dissection Versus Electrocautery Dissection in Endoscopic Nipple-Sparing Mastectomy and Immediate Implant-Based Reconstruction: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-371-02
Record Dates: First submitted 2022-11-30; First posted 2023-09-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms
Keywords: Endoscopy; Mastectomy; Breast Implants; Necrosis; Dissection
MeSH Terms: conditions — Breast Neoplasms; Necrosis

STUDY DESIGN:
Intervention Model Description: Patients who met the inclusion criteria and received informed consent were randomly assigned to the group of using cold separation or the group of using electrocautery with 1:1 allocation based on a computer-generated randomization schedule. The randomization was conducted by drawing an envelope containing the allocation to one of the two intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Dissection (Experimental): In this group, the septa between the skin flap and parenchyma was dissected using with scissors or scalpel
  Interventions: Procedure: Cold dissection
- Electrocautery Dissection (Active Comparator): In this group, the septa between the skin flap and parenchyma was dissected using with electrocautery
  Interventions: Procedure: Electrocautery Dissection

INTERVENTIONS:
Procedure: Cold dissection — The subcutaneous flap dissection was performed with a scissor in this group. The boundary of mastectomy flap was defined as the edge of clavicle superiorly, the edge of sternum medially, the edge of inframammary fold inferiorly, and the edge of the latissimus dorsi laterally. Our tumescent technique utilizes a solution made by mixing 0.2ml of epinephrine with 250 ml of 0.9% Sodium Chloride solution to create a 1‰ ratio. 150ml to 150ml of the solution was injected into the subcutaneous tissue of the operated breast with a 20-gauge spinal needle to establish a bloodless plane. The septa between the skin flap and parenchyma then was dissected using a scissor.
  Arms: Cold Dissection
Procedure: Electrocautery Dissection — The subcutaneous flap dissection was performed with electrocautery in this group. The boundary of mastectomy flap was defined as the edge of clavicle superiorly, the edge of sternum medially, the edge of inframammary fold inferiorly, and the edge of the latissimus dorsi laterally.
  Arms: Electrocautery Dissection

SUMMARY:
The purpose of this study is to analyze whether cold dissection can decrease the rate of ischemia necrosis and other complications and then increase the aesthetic outcomes compared to electrocautery. The purpose of this study is to analyze whether cold dissection can decrease the rate of ischemia necrosis and other complications and then increase the aesthetic outcomes compared to electrocautery.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women in the world. Although breast-conserving surgery is a viable option for patients, mastectomy remains the choice of treatment. Despite oncologic and surgical safety of nipple-sparing mastectomy(NSM) with immediate breast reconstruction(IBR) were amply demonstrated, a number of acute and late complications can occur. Surgical technique may play a role in the postoperative outcomes of mastectomy skin flap.Previous studies suggest that cold dissection with scissors or scalpel, may lead to decreasing blood loss and rates of skin necrosis, compared to electrocautery. A retrospective study by Troy Ng demonstrated that the use of cold dissection is likely to decrease the rate of partial-thickness necrosis (13.0%→33.3%, p=0.01) and full-thickness necrosis (1.3%→12.8%, p=0.02). The purpose of this study is to analyze whether cold dissection can decrease the rate of ischemia necrosis and other complications and then increase the aesthetic outcomes compared to electrocautery.

ELIGIBILITY:
Inclusion Criteria:

* Tumor smaller than 5 cm
* No evidence of NAC, skin or chest wall invasion.
* The general inclusion criteria or pre-requisite for nipple sparing mastectomy apply to E-NSM as well.

Exclusion Criteria:

* Patients with apparent NAC involvement, chest wall or skin invasion, inflammatory breast cancer, locally advanced breast cancer or severe comorbid conditions or poor performance status assessed by the primary physicians, such as heart disease, renal failure, liver dysfunction, and poor performance status as assessed by the primary physicians.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Necrosis complications within one month post operation | Within one month post operation
  Necrosis complications included nipple-areolar complex (NAC) and skin flap necrosis. NAC/skin flap necrosis could present as minor superficial epidermolysis requiring local wound care only, or full-thickness necrosis with any exposure of acellular dermal matrix, muscle, implant, or with full-thickness eschar that required surgical reoperation of debridement and repair.

SECONDARY OUTCOMES:
Necrotic complications within 1 year post operation | Within 1 year post operation
Surgical-site infection rate(SSI) | within one year post operation
  the incidence of surgical-site infection will be compared between two groups
The incidence of postoperative complications | within one year post operation
  the incidence of seroma, hematoma, blister, implant capsular contracture, and implant loss will be compared between two groups
Cosmetic outcomes evaluated by 5-point Likert Scale | Evaluated pre-operation, at the first month, at 2 months, 3 months, 6 months and 12 months.
  Evaluated by patients and five surgeons. In this scale, breast fullness; nipple-areola complex, shape, and contour; scar appearance, size, and fullness; and overall breast appearance will be assessed.
Patient-reported outcomes (as measured using the BREAST-Q score) | Evaluated pre-operation, at the first month, at 2 months, 3 months, 6 months and 12 months.
  The modules included Satisfaction with Breasts, Psychosocial Wellbeing, Sexual Wellbeing, and Physical Wellbeing Chest, Surgeon, Medical Staff, Office Staff.
Postoperative pain | Evaluated at the first day, second day, third day and the first week, second week.
  Pain was assessed using a visual analogue scale(VAS), where 0 = no pain and 10 = worst possible pain.
Total operation time | Immediate post operation
  Defined as the time calculated from the skin incision to the end of wound closure
Intraoperative estimated blood loss | Immediate post operation
  Blood loss (ml) during operation was compared between groups
Drain volume | within three days post operation
  Total drain volume(ml) within three days post operation
Duration of hospital stay post operation | Within 2 weeks of operation.
  Duration of hospital stay post operation(d) will be compared between two group.
Weight of the excised gland | Immediate post operation
  Mean mastectomy weight of patients will be compared between two groups.
Size of implant | Immediate post operation
  Size of implant will be compared between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shicheng Su, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Shicheng Su, Guangzhou, Guangdong, China